CLINICAL TRIAL: NCT02805621
Title: Machine leArning Based CT angiograpHy derIved FFR a Multi-ceNtEr, Registry
Brief Title: Machine leArning Based CT angiograpHy derIved FFR: a Multi-ceNtEr, Registry
Acronym: Machine
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Asan Medical Center (Other); University Hospital, Linkoeping (Other); National Institute of Cardiology, Warsaw, Poland (Other); Medical University of South Carolina (Other); Siemens Healthcare Diagnostics Inc (Industry)
Responsible Party: Principal Investigator, Laurens Groenendijk, dr, Erasmus Medical Center
Other Study IDs: Machine
Record Dates: First submitted 2016-06-15; First posted 2016-06-20 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Coronary Heart Disease; Coronary Artery Disease
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subject: Patients with know or suspected coronary artery disease, who underwent both CT angiography and invasive coronary angiography including invasive FFR measurements.

SUMMARY:
Demonstrate in a large multicenter population the diagnostic performance of a pre-commercial on-site, local, CT angiography derived FFR algorithm in comparison to invasive FFR.

DETAILED DESCRIPTION:
To retrospectively evaluate the diagnostic accuracy of FFRCT, in patients with known or suspected CAD. the investigators propose to do technical assessment of the software and evaluate how different parameters effect the outcome. Validate the FFTCT outcome by comparing the FFRCT values with invasive FFR values from retrospective patient data. To analyze the potential of FFRCT on decision making and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Know or suspect coronary artery disease followed within 6 months by an invasive FFR measurement.

Exclusion Criteria:

* Cardiac event between coronary CT angiography and the invasive FFR procedure, noninterpretable coronary CT angiography image quality, or incomplete coronary CT angiography coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In general, each center used its own specific inclusion and exclusion criteria. Here the investigators describe the general criteria, please see the respected publications for a detailed description.1-4
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2016-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of local reduced order CFD and machine learning based CT angiography derived FFR, both validated against invasive FFR. Measured at both vessel and patient level. | 6 months

SECONDARY OUTCOMES:
Influence of calcium on diagnostic accuracy of CT angiography derived FFR. | 6 months
Confidence intervals of CT angiography derived FFR | 6 months
Direct vessel based comparison between CT angiography derived FFR and QCT stenosis measurements | 6 months
Analysis of anatomically mild stenosis (<50% lumen diameter reduction) but functionally significant (invasive FFR ≤ 0.80) | 6 months
Long term clinical outcome of CT angiography derived FFR | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Koen Nieman, MD PHD, Principal Investigator — Erasmus Medical Center
Locations (1):
- ErasmusMC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Geer J, Sandstedt M, Bjorkholm A, Alfredsson J, Janzon M, Engvall J, Persson A. Software-based on-site estimation of fractional flow reserve using standard coronary CT angiography data. Acta Radiol. 2016 Oct;57(10):1186-92. doi: 10.1177/0284185115622075. Epub 2015 Dec 20. PMID 26691914
- [Background] Kruk M, Wardziak L, Demkow M, Pleban W, Pregowski J, Dzielinska Z, Witulski M, Witkowski A, Ruzyllo W, Kepka C. Workstation-Based Calculation of CTA-Based FFR for Intermediate Stenosis. JACC Cardiovasc Imaging. 2016 Jun;9(6):690-9. doi: 10.1016/j.jcmg.2015.09.019. Epub 2016 Feb 17. PMID 26897667
- [Background] Baumann S, Wang R, Schoepf UJ, Steinberg DH, Spearman JV, Bayer RR 2nd, Hamm CW, Renker M. Coronary CT angiography-derived fractional flow reserve correlated with invasive fractional flow reserve measurements--initial experience with a novel physician-driven algorithm. Eur Radiol. 2015 Apr;25(4):1201-7. doi: 10.1007/s00330-014-3482-5. Epub 2014 Nov 18. PMID 25403173
- [Background] Coenen A, Lubbers MM, Kurata A, Kono A, Dedic A, Chelu RG, Dijkshoorn ML, Gijsen FJ, Ouhlous M, van Geuns RJ, Nieman K. Fractional flow reserve computed from noninvasive CT angiography data: diagnostic performance of an on-site clinician-operated computational fluid dynamics algorithm. Radiology. 2015 Mar;274(3):674-83. doi: 10.1148/radiol.14140992. Epub 2014 Oct 13. PMID 25322342
- [Background] Yang DH, Kim YH, Roh JH, Kang JW, Ahn JM, Kweon J, Lee JB, Choi SH, Shin ES, Park DW, Kang SJ, Lee SW, Lee CW, Park SW, Park SJ, Lim TH. Diagnostic performance of on-site CT-derived fractional flow reserve versus CT perfusion. Eur Heart J Cardiovasc Imaging. 2017 Apr 1;18(4):432-440. doi: 10.1093/ehjci/jew094. PMID 27354345
- [Derived] Tesche C, Otani K, De Cecco CN, Coenen A, De Geer J, Kruk M, Kim YH, Albrecht MH, Baumann S, Renker M, Bayer RR, Duguay TM, Litwin SE, Varga-Szemes A, Steinberg DH, Yang DH, Kepka C, Persson A, Nieman K, Schoepf UJ. Influence of Coronary Calcium on Diagnostic Performance of Machine Learning CT-FFR: Results From MACHINE Registry. JACC Cardiovasc Imaging. 2020 Mar;13(3):760-770. doi: 10.1016/j.jcmg.2019.06.027. Epub 2019 Aug 14. PMID 31422141